CLINICAL TRIAL: NCT02093468
Title: Evaluation of MST-188 in Acute Lower Limb Ischemia: A Phase 2 Randomized, Double-Blind, Placebo-Controlled, Multi-Center Clinical Trial Evaluating the Safety and Efficacy of MST-188 in Subjects With Acute Lower Limb Ischemia Receiving Catheter-Directed Recombinant Tissue Plasminogen Activator
Brief Title: Evaluation of MST-188 in Acute Lower Limb Ischemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Program discontinued to persue alternate indications.
Sponsor: Mast Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MST-188-07
Record Dates: First submitted 2014-03-18; First posted 2014-03-21 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Acute Limb Ischemia
Keywords: Acute limb ischemia; ALI; Acute lower extremity arterial occlusion
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Saline (Placebo Comparator): Saline administered IV for 12 hours
  Interventions: Drug: Saline
- Lower Dose (Experimental): MST-188 loading dose 100 mg/kg IV for 1 hour followed by 25 mg/kg/hr for 11 hours
  Interventions: Drug: MST-188
- Higher Dose (Experimental): MST-188 loading dose 200 mg/kg IV for 1 hour followed by 75 mg/kg/hr for 11 hours
  Interventions: Drug: MST-188

INTERVENTIONS:
Drug: MST-188
  Other Names: vepoloxamer
  Arms: Higher Dose; Lower Dose
Drug: Saline
  Arms: Saline

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of MST-188 in subjects receiving catheter-directed rt-PA for acute lower limb ischemia and to evaluate whether treatment with MST-188 results in more rapid thrombolysis of the occlusion and more rapid tissue perfusion in the effected blood vessel.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥30 to <80
* Symptoms consistent with ALI in target lower limb classified as Rutherford Category IIa or IIb
* Subject is hospitalized or in the process of hospitalization for the treatment of ALI
* Angiographic confirmation of thrombotic lower limb arterial occlusion

Exclusion Criteria:

* Prosthetic bypass graft occlusion within 1 month of implantation or autogenous graft occlusion within 6 months of placement
* Treatment with a thrombolytic agent within the last 48 hours
* Subject's laboratory results indicate inadequate organ function
* NYHA Class IV congestive heart failure
* Prior major amputation of the target limb
* Other complications or contraindications for receiving rt-PA, anticoagulants, or contrast media

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-06; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Angiographic assessment of the change in the volume of thrombus (Exploratory endpoint) | Baseline, 8 and 24 hours
Assessment of the change in TcPO2 (Exploratory endpoint) | Baseline, 8, 12, and 24 hours
Number of participants with adverse events | Randomization through 30 days post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Edwin L Parsley, D.O., Study Director — Mast Therapeutics, Inc.
Locations (4):
- United States (4):
  - Research Center, Little Rock, Arkansas
  - Research Center, Tampa, Florida
  - Research Center, Brooklyn, New York
  - Research Center, Cleveland, Ohio